CLINICAL TRIAL: NCT03964493
Title: Phase 2, Double-Blind, Randomized, Multicenter, Parallel, Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of TNP-2092 to Treat Acute Bacterial Skin and Skin Structure Infection in Adults
Brief Title: TNP-2092 to Treat Acute Bacterial Skin and Skin Structure Infection
Acronym: P2_ABSSSI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TenNor Therapeutics Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PJI001-02
Record Dates: First submitted 2019-04-30; First posted 2019-05-28 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections; Gram-Positive Bacterial Infections
Keywords: TNP-2092; ABSSSI; Safety; Efficacy
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — TNP-2092; Vancomycin

STUDY DESIGN:
Intervention Model Description: TNP-2092 300 mg intravenous every 12 hours vancomycin 1 g intravenous every 12 hours
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNP-2092 (Experimental): TNP-2092 300 mg intravenous every 12 hours
  Interventions: Drug: TNP-2092
- Vancomycin (Active Comparator): vancomycin 1 g intravenous every 12 hours
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: TNP-2092 — TNP-2092 100mg/vial
  Arms: TNP-2092
Drug: Vancomycin — Vancomycin 1g/vial
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetic characteristics and efficacy of TNP-2092 in adults with ABSSSI suspected or confirmed to be caused by gram-positive pathogens.

DETAILED DESCRIPTION:
This Phase 2, double-blind, randomized, multicenter, parallel, controlled study is conducted to evaluate safety, tolerability, pharmacokinetics and efficacy of TNP-2092, and vancomycin in adults with ABSSSI suspected or confirmed to be caused by gram-positive pathogens. The duration of the treatment period is a minimum of 7 days and a maximum of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included in the study if they meet all of the following inclusion criteria:

  * Males or females, 18 years of age or older;
  * ABSSSI suspected or confirmed to be caused by gram-positive pathogens, including:
  * Cellulitis/erysipelas;
  * Wound infection;
  * Major cutaneous abscess;
  * Lesion with a minimum surface area of 75 cm2;
  * Capable of giving signed informed consent.

Exclusion Criteria:

* Subjects will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

  * History or hypersensitivity or intolerability to any fluoroquinolone, rifamycin or glycopeptide classes;
  * ABSSSI suspected or confirmed to be caused by pathogens that are resistant to the glycopeptide class;
  * Prior administration of systemic antibacterial therapy within 96 hours before randomization;
  * ABSSSI with suspected or confirmed infection caused by gram-negative or anaerobic organisms;
  * ABSSSI with suspected or confirmed infection caused by fungal, mycobacterial, parasitic, or viral pathogens;
  * Evidence of significant hepatic, hematologic, or immunologic disease;
  * History or evidence of severe renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TenNor Clinical Trials, Study Director — TenNor
Locations (1):
- eStudy Site, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNP-2092 | Vancomycin
Started | 80 | 40
Completed | 63 | 35
Not Completed | 17 | 5
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNP-2092 | Vancomycin | Total
Number analyzed (Participants) | 80 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.72) | 42.7 (13.16) | 41.9 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 61 | 26 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 17 | 49
  Not Hispanic or Latino | 48 | 23 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 70 | 32 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Height [Mean (Standard Deviation); unit: cm] | 173.5 (9.46) | 170.5 (8.32) | 172.5 (9.17)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (2.98) | 24.8 (3.47) | 24.4 (3.15)
Weight [Mean (Standard Deviation); unit: kg] | 72.8 (11.81) | 72.7 (14.43) | 72.8 (12.68)

OUTCOME MEASURES:

1. Primary Outcome: Early Clinical Response at the Early Assessment (EA) Visit in the Intent-to-Treat (ITT) Population
Description: Early clinical response is defined as responder meeting two criteria: (1) patient had at least a 20% reduction of acute bacterial skin and skin structure infection (ABSSSI) primary lesion size compared to baseline measurements; (2) patient did not die of any cause within 72 hours of the first dose of study treatment. An indeterminate classification is used for a response that could not be adequately inferred because study data are unavailable for evaluation of efficacy for any reason (eg, missing data, lost to follow-up, did not attend the EA clinic appointment), or if the early assessment visit is out of the 48 to 72 hours window after the intravenous study treatment starts.
Time Frame: 48 to 72 hours after the first dose of study treatment
Population: Intent-to-Treat (mITT) Population: all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 80 | 40
Participants
  Responder | 61 | 27
  Nonresponder | 4 | 3
  Indeterminate | 15 | 10

2. Primary Outcome: Early Clinical Response at the Early Assessment Visit in the Modified Intent-to-Treat (mITT) Population
Description: as for outcome 1
Time Frame: 48 to 72 hours after the first dose of study treatment
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants in the ITT population excluding those who have gram-negative pathogens only
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 78 | 40
Participants
  Responder | 60 | 27
  Nonresponder | 4 | 3
  Indeterminate | 14 | 10

3. Primary Outcome: Early Clinical Response at the Early Assessment Visit in the Micro-Intent-to-Treat (Micro-ITT) Population
Description: as for outcome 1
Time Frame: 48 to 72 hours after the first dose of study treatment
Population: Micro-Intent-to-Treat (mITT) Population: all randomized participants in the mITT population with culture evidence of a baseline gram-positive ABSSSI pathogens (exclude sole gram negative and culture-negative participants)
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 51 | 29
Participants
  Responder | 41 | 19
  Nonresponder | 3 | 2
  Indeterminate | 7 | 8

4. Secondary Outcome: Investigator Assessment of Clinical Response at Post Treatment Evaluation (PTE) Visit in the mITT Population
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; the ABSSSI sufficiently resolved such that further antibacterial therapy is not needed. Clinical Failure: any of the following: (1)Investigator discontinued study treatment and indicated that the ABSSSI had responded inadequately such that alternative (rescue) non-study antibacterial therapy was needed; (2)participant received antibacterial therapy for a different infection that may be effective for the ABSSSI under study; (3) participant developed an adverse event (AE) that required discontinuation of study treatment before completion of the planned treatment regimen; (4) unplanned major surgical treatment for the ABSSSI under study; (5) participant died of any cause up to the specified visit. Indeterminate: study data are unavailable for evaluation of efficacy for any reason (eg, missing data, lost to follow-up).
Time Frame: 7 to 14 days after the end of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 78 | 40
Participants
  Success | 62 | 31
  Failure | 2 | 3
  Indeterminate | 14 | 6

5. Secondary Outcome: Investigator Assessment of Clinical Response at Post Treatment Evaluation (PTE) Visit in the Micro-ITT Population
Description: as for outcome 4
Time Frame: 7 to 14 days after the end of study treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 51 | 29
Participants
  Success | 40 | 23
  Failure | 2 | 1
  Indeterminate | 9 | 5

6. Secondary Outcome: Investigator's Assessment of Clinical Response at the End of Treatment (EOT) Visit in the mITT Population
Description: At the EOT Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; the ABSSSI sufficiently resolved such that further antibacterial therapy is not needed. Clinical Failure: any of the following: (1)Investigator discontinued study treatment and indicated that the ABSSSI had responded inadequately such that alternative (rescue) non-study antibacterial therapy was needed; (2)participant received antibacterial therapy for a different infection that may be effective for the ABSSSI under study; (3) participant developed an adverse event (AE) that required discontinuation of study treatment before completion of the planned treatment regimen; (4) unplanned major surgical treatment for the ABSSSI under study; (5) participant died of any cause up to the specified visit. Indeterminate: study data are unavailable for evaluation of efficacy for any reason (eg, missing data, lost to follow-up).
Time Frame: After a minimum of 7 days up to 14 days of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 78 | 40
Participants
  Success | 68 | 31
  Failure | 2 | 3
  Indeterminate | 8 | 6

7. Secondary Outcome: Investigator's Assessment of Clinical Response at the End of Treatment (EOT) Visit in the Micro-ITT Population
Description: as for outcome 6
Time Frame: After a minimum of 7 days up to 14 days of study treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TNP-2092 | Vancomycin
Number analyzed (Participants) | 51 | 29
Participants
  Success | 45 | 23
  Failure | 2 | 1
  Indeterminate | 4 | 5

8. Secondary Outcome: AUC0-12h After First Infusion
Description: Partial area under the concentration versus time curve from time zero to time 12 hours.
Time Frame: 0 to 12 hours post-dose
Population: Participants that have sufficient plasma points for AUC 0-12h after first infusion analysis (26 Participants).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNP-2092
Number analyzed (Participants) | 26
h*ng/mL | 135000 (38200)

9. Secondary Outcome: AUC0-12h After Last Infusion
Description: Partial area under the concentration versus time curve from time zero to time 12 hours
Time Frame: 0 to 12 hours post-dose
Population: Participants that have sufficient plasma points for AUC 0-12h after last infusion analysis (39 Participants)
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TNP-2092
Number analyzed (Participants) | 39
h*ng/mL | 159000 (74200)

10. Secondary Outcome: Cmax After Last Infusion
Description: Maximum observed concentration
Time Frame: 57 to 60 minutes, 1.5 to 3 hours, 4 to 6 hours, 12 hours, after the last infusion
Population: Participants that have sufficient plasma points for Cmax after last infusion analysis (58 Participants)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TNP-2092
Number analyzed (Participants) | 58
ng/mL | 38500 (13400)

11. Secondary Outcome: Cmax After First Infusion
Description: Maximum observed concentration
Time Frame: 57 to 60 minutes, 1.5 to 3 hours, 4 to 6 hours, 12 hours, after the first infusion
Population: Participants that have sufficient plasma points for Cmax after first infusion analysis (68 Participants)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TNP-2092
Number analyzed (Participants) | 68
ng/mL | 37500 (13500)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the first day of study treatment (day 1) to long-term follow-up visit(20 to 25 days after end of treatment), A Serious Adverse event (SAE) will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up.
Description: Adverse events are reported for members of the Safety Population, comprised of all randomized participants who received any amount of study treatment. Treatment-emergent adverse events, defined as events occurring after initiation of study treatment, are reported.
Arm/Group | TNP-2092 | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/78 | 2/39
Other Adverse Events (participants affected / at risk) | 27/78 | 11/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 (N=78) | Vancomycin (N=39)
MRSA bacteremia and worsening cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant 002-0071 (TNP-2092 group) had a severe serious adverse event (SAE) of staphylococcal infection (MRSA bacteremia and worsening cellulitis) on Day 2, considered unrelated to study treatment and the SAE recovered on Day 8.
mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) — Participant 002-0038 in the vancomycin group had a moderate SAE of mental status changes related to opioid overdose on Day 18. The SAE was considered unrelated to study treatment and the SAE recovered/resolved on Day 19.
left upper extremity abscess,dehydration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Participant 003-0031 in the vancomycin group had 2 SAEs: A severe SAE of left upper extremity abscess on Day 4. A severe SAE of dehydration on Day 47. The SAEs were considered unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 (N=78) | Vancomycin (N=39)
Nausea (Gastrointestinal disorders) | 12 (12) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Wound infection (Infections and infestations) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03964493/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03964493/SAP_003.pdf